CLINICAL TRIAL: NCT00260039
Title: A Randomized, International, Double-Blinded (With In-House Blinding), GARDASIL-Controlled, Dose-Ranging Study of Octavalent Human Papillomavirus (HPV) L1 Virus-like Particle (VLP) Vaccine Administered to 16- to 23- Year-Old Women
Brief Title: Broad Spectrum HPV Vaccine Dose Ranging Study (V502-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V502-001; 2005_086
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: HPV; Cervical Cancer; Premalignancy Anogenital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Active Comparator): Gardasil
  Interventions: Biological: Comparator: Gardasil
- 2 (Experimental): HPV VLP vaccine -Dose regimen 1
  Interventions: Biological: Comparator: octavalent HPV Vaccine - dose formulation 1
- 3 (Experimental): HPV VLP vaccine -Dose regimen 2
  Interventions: Biological: Comparator: octavalent HPV Vaccine - dose formulation 2
- 4 (Experimental): HPV VLP vaccine -Dose regimen 3
  Interventions: Biological: Comparator: octavalent HPV Vaccine - dose formulation 3

INTERVENTIONS:
Biological: Comparator: Gardasil — 0.5 mL intramuscular injection administered at Day 1, Month 2 and Month 6
  Arms: 1
Biological: Comparator: octavalent HPV Vaccine - dose formulation 1 — 0.5 mL octavalent HPV vaccine - intramuscular injection administered at Day 1, Month 2 and Month 6
  Arms: 2
Biological: Comparator: octavalent HPV Vaccine - dose formulation 2 — 0.5 mL octavalent HPV vaccine - intramuscular injection administered at Day 1, Month 2 and Month 6
  Arms: 3
Biological: Comparator: octavalent HPV Vaccine - dose formulation 3 — 0.5 mL octavalent HPV vaccine - intramuscular injection administered at Day 1, Month 2 and Month 6
  Arms: 4

SUMMARY:
This dose-ranging study is to evaluate an investigational vaccine with the following objectives: (1) To demonstrate that the vaccine is well-tolerated in women (2) To evaluate immune responses in women who are between 16 and 23 years of age at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime history of 0-4 sexual partners

Exclusion Criteria:

* History of abnormal PAP test or abnormal cervical biopsy result; history of external genital/vaginal warts; history of positive HPV test

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 680 (Actual)
Dates: Start 2005-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The octavalent HPV VLP vaccine, when administered in a 3-dose regimen, induces acceptable responses for specific HPV types at 4 weeks Post dose 3. Immune responses measured by an HPV competitive Luminex immunoassay. | 4 weeks post dose 3 injection

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Luxembourg A, Brown D, Bouchard C, Giuliano AR, Iversen OE, Joura EA, Penny ME, Restrepo JA, Romaguera J, Maansson R, Moeller E, Ritter M, Chen J. Phase II studies to select the formulation of a multivalent HPV L1 virus-like particle (VLP) vaccine. Hum Vaccin Immunother. 2015;11(6):1313-22. doi: 10.1080/21645515.2015.1012010. PMID 25912208